CLINICAL TRIAL: NCT00980083
Title: Endogenous GLP-1 Regulates Postprandial Glycaemia in Human: Relative Contributions of Insulin, Glucagon, and Gastric Emptying
Brief Title: GLP-1 - Regulatory Mechanism of Postprandial Glycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: University of Munich
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MSE
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects; Gastric Emptying
Keywords: GLP-1; exendin(9-39); gastric emptying; incretin; human
MeSH Terms: interventions — Sodium Chloride; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline
- Exendin(9-39) (Active Comparator)
  Interventions: Drug: Exendin(9-39)amide

INTERVENTIONS:
Drug: Saline
  Arms: Placebo
Drug: Exendin(9-39)amide
  Arms: Exendin(9-39)

SUMMARY:
Synthetic GLP-1 lowers postprandial (pp) glycemia by stimulating insulin, inhibiting glucagon, and delaying gastric emptying. However, the effects of the endogenous peptide are largely unknown. Using the specific GLP-1 receptor antagonist exendin(9-39)amide (Ex(9-39)) the investigators recently showed that GLP-1 released during intestinal meal perfusion acts as an incretin hormone and as an enterogastrone. As the relative contributions of these effects to controll postprandial glycemia are unclear, the investigators used Ex(9-39) to investigate the mechanisms of action of GLP-1 after an oral meal in humans.

DETAILED DESCRIPTION:
Two experiments were performed in random order in 12 healthy subjects. After a 50-min basal period subjects ingested a 412 kcal mixed semisolid meal containing 30g oatmeal, labelled with 99mTc-Sn-colloid. Gastric emptying was measured by high-resolution scintigraphy until 210 min after meal ingestion. Saline (SAL) or Ex(9-39) at 900 pmol/kg/min was intravenously infused during the two experiments. In addition, in 6 of the 12 subjects gastric motility was measured by antroduodenal manometry and gastric barostat. AUC: pp incremental area under the curve. Lag period (LP): time to 10% emptying.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* >=18 years of age
* No medication

Exclusion Criteria:

* Acute disease
* Metabolic disease
* On medication
* Pregnancy, breast feeding
* Gastrointestinal surgery
* Dyspeptische Symptome (Völlegefühl, Blähungen, abdominelle Schmerzereignisse, Übelkeit, Erbrechen, Sodbrennen)
* Teilnahme an einer klinischen Studie in den vergangenen 6 Monaten

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-10; Primary Completion 2005-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
postprandial blood glucose levels | -50 min until 210 min after meal intake

SECONDARY OUTCOMES:
gastric emptying rate | 0-210min
plasma levels of glucagon, insulin | -50min until 210 min

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, Prof, Principal Investigator — University of Munich, Department of Internal Medicine II, Munich, Germany
Locations (1):
- Department of Internal Medicine II, University of Munich, Munich, Germany